CLINICAL TRIAL: NCT02075463
Title: A 16-week, Phase 2a, Single-arm, Multi-center, Open-label Study to Evaluate the Safety and Efficacy of GSK1278863 After Switching From Recombinant Human Erythropoietin (rhEPO), in Hemodialysis-dependent Subjects With Anemia Associated With Chronic Kidney Disease Who Are Chronically Hyporesponsive to rhEPO
Brief Title: Study to Evaluate the Safety and Efficacy of GSK1278863 in Recombinant Human Erythropoietin (rhEPO) Hyporesponsive Hemodialysis-dependent Chronic Kidney Disease Subjects With Anemia
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 114837
Record Dates: First submitted 2014-02-27; First posted 2014-03-03 (Estimated); Results first posted 2017-06-21 (Actual); Last update posted 2017-06-21 (Actual); Status verified 2017-04

CONDITIONS: Anemia
Keywords: recombinant human erythropoietin; GSK1278863; hemodialysis; anemia; Hemoglobin; chronic rhEPO hyporesponsiveness; chronic kidney disease; erythropoiesis stimulating agents; pharmacokinetics
MeSH Terms: conditions — Anemia; Renal Insufficiency, Chronic | interventions — GSK1278863

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- GSK1278863 Arm (Experimental): Subjects will receive a fixed starting dose of 12 milligrams (mg) GSK1278863 once daily (QD) orally for first 4 weeks. From Week 4 the dose of GSK1278863 will be adjusted based on Hgb levels and evaluated every 4 weeks until Week 16. This starting dose may be changed during the study if there is an early indication of either lack of efficacy or the rate of rise in Hgb is too rapid
  Interventions: Drug: GSK1278863; Drug: Placebo

INTERVENTIONS:
Drug: GSK1278863 — Film coated tablets containing 1 mg, 2 mg, 5 mg or 25 mg of GSK1278863
Drug: Placebo — Matching placebo tablet for GSK1278863

SUMMARY:
The study will evaluate the ability of GSK1278863 to increase the hemoglobin (Hgb) concentration, or maintain it within the target range, and the safety and efficacy of GSK1278863 over 16 weeks of treatment, in hemodialysis-dependent subjects with anemia associated with chronic kidney disease who are chronically hyporesponsive to rhEPO. The data generated will inform dose requirements for any chronic rhEPO hyporesponsive hemodialysis-dependent subjects included in future clinical trials. The study consists of a 4-week rhEPO run-in period, a 16-week GSK1278863 treatment period and a 4-week Follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* Hemodialysis (HD) frequency: Stable HD regimen of three to four times weekly for a minimum of 12 weeks. Note: The type and frequency of dialysis must be stable during the study. Isolated ultrafiltration sessions for the purposes of fluid removal are permitted.
* Dialysis Adequacy: Single-pool dialyzer clearance multiplied by dialyzer time divided by volume of distribution of urea (Kt/Vurea) of >=1.2 based on a historical value obtained within the prior month.
* rhEPO hyporesponsiveness: Historical and current intravenous (IV) rhEPO and Hgb values. Average epoetin alfa dose and Hgb level for three 4-week periods for a total of 12 weeks prior to Week -4, and during the 4 week run-in period, must be within the following ranges: average epoetin alfa dose >4000 and <=6000 units per session and Hgb >=8.0 and <=9.5 g/dL; average epoetin alfa dose >6000 and <=8000 units per session and Hgb >=8.0 and <=10.0 g/dL; average epoetin alfa dose >8000 and <=10000 units per session and Hgb >=8.0 and <=10.5 g/dL; and average epoetin alfa dose >10000 units per session and Hgb >=8.0 and <=11.0 g/dL.
* Absolute difference between the Hgb value at Week -4 and Week 0 (Day 1), must be <1.3 g/dL. Note: Subjects who do not meet the criteria after being rescreened twice, should not be entered into the GSK1278863 treatment period and should be withdrawn from the study.
* Age: >=18 years of age.
* Q-T Interval Corrected for Heart Rate (QTc): Bazett's Correction of QT Interval (QTcB) <470 msec or QTcB <480 milliseconds (msec) in subjects with bundle branch block. There is no corrected QT interval (QTc) inclusion criterion for a subject with a predominantly paced rhythm.
* Gender: Female and male subjects. Females: If of childbearing potential, must agree to use one of the approved contraception methods from Screening until completion of the Follow-up Visit OR, of non-childbearing potential defined as pre-menopausal females with a documented tubal ligation, hysterectomy or oophorectomy; or postmenopausal defined as 12 months of spontaneous amenorrea [in questionable cases a blood sample with simultaneous follicle stimulating hormone (FSH) 23.0-116.3 milliinternational units (MIU)/milliliter (mL) (23.0-116.3 international units (IU)/liter (L)) and estradiol <=10 picograms (pg)/mL (<=37 picomole (pmol)/L) is confirmatory]. Females on hormone replacement therapy (HRT) whose menopausal status is in doubt will be required to use one of the approved contraception methods if they wish to continue their HRT during the study. Otherwise they must discontinue HRT to allow confirmation of post-menopausal status prior to study enrollment. For most forms of HRT, at least 2 weeks will elapse between the cessation of therapy and the blood draw; this interval depends on the type and dosage of HRT. Following confirmation of their post-menopausal status, they can resume use of HRT during the study without use of a contraceptive method.

Exclusion Criteria:

* Dialysis modality: Planned change in dialysis modality within the study time period.
* rhEPO: Use of methoxy polyethylene glycol epoetin beta or darbepoetin within the prior 8 weeks prior to Week -4.
* Renal transplant: Scheduled renal transplant.
* Transferrin saturation (TSAT): <20% on the most recent sample taken over the last 12 weeks.
* Ferritin: <100 nanograms (ng)/mL (<100 micrograms/L) on the most recent sample taken over the last 12 weeks.
* Vitamin B12: At or below the lower limit of the reference range (may rescreen in a minimum of 8 weeks).
* Folate: <2.0 ng/mL (<4.5 nanomoles (nmol)/L) (may rescreen in a minimum of 4 weeks).
* Myocardial infarction or acute coronary syndrome: Within the 8 weeks prior to Week -4.
* Stroke or transient ischemic attacks (TIAs): Within the 8 weeks prior to Week -4.
* Heart failure: Class III/IV heart failure, as defined by the New York Heart Association (NYHA) functional classification system diagnosed prior to Week -4.
* Hypertension: Defined using pre-dialysis vitals (Week -4) of diastolic blood pressure >100 millimeters of mercury (mmHg) or systolic blood pressure >170 mmHg.
* Thrombotic disease: History of thrombotic disease (e.g., venous thrombosis such as deep vein thrombosis or pulmonary embolism, or arterial thrombosis such as new onset or worsening limb ischemia requiring intervention) within the 8 weeks prior to Week -4, except vascular access thrombosis.
* Inflammatory disease: Active chronic inflammatory disease that could impact erythropoiesis (e.g., scleroderma, systemic lupus erythematosis, rheumatoid arthritis, celiac disease) diagnosed prior to Week -4.
* Hematological disease: Any hematological disease including those affecting platelets, white or red blood cells (e.g., antibody-mediated pure red cell aplasia, sickle cell anemia, myelodysplastic syndromes, hematological malignancy, myeloma, hemolytic anemia), coagulation disorders (e.g., antiphospholipid syndrome, Protein C or S deficiency), or any other cause of anemia other than renal disease diagnosed prior to Week -4.
* Liver disease: Current liver disease, known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones) or evidence at Screening of abnormal liver function tests [alanine transaminase (ALT) or aspartate transaminase (AST) > 2.0 x upper limit of normal (ULN) or total bilirubin > 1.5 x ULN]; or other hepatic abnormalities that in the opinion of the investigator would preclude the subject from participation in the study. NOTE: Those with Hepatitis B or Hepatitis C are eligible provided these exclusions are not met.
* Major surgery: (excluding vascular access surgery) within the 8 weeks prior to Week -4, or planned during the study.
* Transfusion: Blood transfusion within the 8 weeks prior to Week -4, or an anticipated need for blood transfusion during the study.
* Gastrointestinal (GI) Bleeding: Evidence of actively bleeding peptic, duodenal, or esophageal ulcer disease or clinically significant GI bleeding within the 8 weeks prior to Week -4.
* Ophthalmology disease: History of proliferative retinopathy requiring treatment within the prior 12 months or macular edema requiring treatment.
* Acute infection: Clinical evidence of acute infection, evidence of underlying infection or history of infection requiring IV antibiotic therapy within the 8 weeks prior to Week -4, and also through to Day 1. Note: IV antibiotics as prophylaxis are allowed.
* Malignancy: Subjects with a history of malignancy within the prior 5 years, who are receiving treatment for cancer, or who have a strong family history of cancer (e.g., familial cancer disorders), with the exception of squamous cell or basal cell carcinoma of the skin that has been definitively treated prior to Week -4.
* Severe allergic reactions: History of severe allergic or anaphylactic reactions or hypersensitivity to excipients in the investigational product.
* Drugs and supplements: Use of any prescription or non-prescription drugs or dietary supplements that are prohibited from Week -4 until the Follow-up Visit.
* Prior investigational product exposure: The subject has participated in a clinical trial and has received an experimental investigational product within the prior 30 days to Week -4.
* Life Expectancy: Life expectancy is considered by the investigator to be less than 6 months.
* Other conditions: Any other conditions, clinical or laboratory abnormality, or examination finding that the Investigator considers would put the subject at unacceptable risk, or an unwillingness or inability to follow the procedures, or lifestyle and/or dietary restrictions outlined in the protocol.
* Pregnancy and lactation: Pregnant females as determined by positive serum human chorionic gonadotrophin (hCG) test or women who are lactating at Week -4 or during the trial.
* Laboratory eligibility criteria will be assessed according to the central laboratory result for the screening samples
* Subjects who fail screening may be rescreened as soon as the investigator feels they may have subsequently become eligible. However, an individual subject may not be rescreened more than twice. There is no predetermined amount of time required to wait to rescreen a previously ineligible subject. Exceptions are those failing on Hgb or folate who may rescreen in 4 weeks and those failing for Vitamin B12 where rescreening may occur in 8 weeks.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2014-06-01; Primary Completion 2016-03-01 (Actual); Study Completion 2016-03-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (18):
- United States (18):
  - GSK Investigational Site, Azusa, California
  - GSK Investigational Site, Glendale, California
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, Paramount, California
  - GSK Investigational Site, San Diego, California
  - GSK Investigational Site, Simi Valley, California
  - GSK Investigational Site, Middlebury, Connecticut
  - GSK Investigational Site, Hollywood, Florida
  - GSK Investigational Site, Tampa, Florida
  - GSK Investigational Site, Macon, Georgia
  - GSK Investigational Site, Southgate, Michigan
  - GSK Investigational Site, Saint Ann, Missouri
  - GSK Investigational Site, St Louis, Missouri
  - GSK Investigational Site, Amherst, New York
  - GSK Investigational Site, Asheville, North Carolina
  - GSK Investigational Site, Bethlehem, Pennsylvania
  - GSK Investigational Site, Knoxville, Tennessee
  - GSK Investigational Site, Houston, Texas

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Eligible hemodialysis-dependent participants (par.) with anemia associated with chronic kidney disease and chronically hyporesponsive to recombinant human erythropoietin (rhEPO) (for 12 weeks) were switched from a stable dose of rhEPO
Pre-assignment Details: Study consisted of run-in period of 4 weeks (wk), 16-wk Treatment Phase and Follow-up period of 4-wk after completion of treatment.
Groups:
- GSK1278863 12 mg QD: Participants received a fixed dose GSK1278863 12 milligram (mg) once daily (QD) for the first 4 weeks. After Week 4, the dose was adjusted every four weeks to achieve hemoglobin (Hgb) levels within the range of 10.0-11.5 grams (g)/deciliter (dL); however, a dose decrease was also permitted for a subject at Week 2 if the rise in Hgb is too rapid.
Period: Overall Study
Arm/Group | GSK1278863 12 mg QD
Started | 15
Completed | 7
Not Completed | 8
Not completed — Adverse Event | 3
Not completed — Par. reached stopping criteria | 4
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | GSK1278863 12 mg QD
Number analyzed (Participants) | 15
Age, Continuous [Mean (Standard Deviation); unit: Years] | 59.1 (12.76)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 8
Race/Ethnicity, Customized [Number; unit: Participants]
  BLACK OR AFRICAN AMERICAN | 2
  WHITE | 13

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Demonstrating an Increase in Hgb of >=1 g/dL (if Baseline Hgb is <9.5 g/dL), or >=0.5 g/dL (if Baseline Hgb is 9.5-<10 g/dL), or Stay Within Target Range and do Not Drop by >0.5 g/dL (if Baseline Hgb is >= 10 g/dL) at Week 16
Description: Percentage of participants with increased Hgb >=1 g/dL (if baseline Hgb is <9.5 g/dL), or >=0.5 g/dL (if baseline Hgb is 9.5-<10 g/dL), or within the target range and not dropped by >0.5 g/dL (if baseline Hgb is >= 10 g/dL) at Week 16 are presented. Participants who were available at the indicated time point were analyzed
Time Frame: Week 16
Population: ITT population: participants who received at least one dose of drug, have a baseline Hgb and at least one corresponding on treatment Hgb assessment.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | GSK1278863 12 mg QD
Number analyzed (Participants) | 7
Percentage of participants | 28.6 [8.2 to 64.1]

2. Secondary Outcome: Change From Baseline in Hgb Levels at Week 16
Description: Hgb values measured at Week 16 are presented. Change from baseline was calculated as Week 16 minus baseline value . Participants who were available at the indicated time point were analyzed.
Time Frame: Week 16
Population: ITT population.
Measure: Mean (Standard Deviation); unit: g/dL
Groups:
- GSK1278863 12 mg QD: Participants received a fixed dose GSK1278863 12 mg QD for the first 4 weeks. After Week 4, the dose was adjusted every four weeks to achieve Hgb levels within the range of 10.0-11.5 g/dL; however, a dose decrease was also permitted for a subject at Week 2 if the rise in Hgb is too rapid.
Arm/Group | GSK1278863 12 mg QD
Number analyzed (Participants) | 7
g/dL | 0.10 (1.319)

3. Secondary Outcome: Percentage of Time (Days) Hgb Levels Within, Below and Above Target Range at the Indicated Time Point
Description: The percentage of time in Hgb levels were in target range (10.0 to 11.5 g/dL) between Weeks 12 and 16 for a participant was calculated by adding the total number of days that Hgb is within target range while on treatment during Weeks 12 to 16 and dividing by the total number of days the participant remained on treatment during Weeks 12 to 16 (using Rosendaal linear interpolation method). Similarly, percentage of time above Hgb target range and percentage of time below Hgb target range were calculated. Participants who were available at the indicated time point were analyzed.
Time Frame: Week 12 to Week 16
Population: ITT population.
Measure: Mean (Standard Deviation); unit: Percentage of days
Arm/Group | GSK1278863 12 mg QD
Number analyzed (Participants) | 8
Percentage of days
  Within Target Range | 48.28 (46.102)
  Above target range | 0.92 (2.605)
  Below target range | 50.80 (47.176)

4. Secondary Outcome: Number of Participants Achieving at Least 1 g/dL Increase in Hgb From Baseline at Week 16
Description: Number of participants achieving at least 1 g/dL increase in Hgb from baseline at Week 16 were presented. Participants who were available at the indicated time point were analyzed.
Time Frame: Baseline and Week 16
Population: ITT population.
Measure: Number; unit: Participants
Arm/Group | GSK1278863 12 mg QD
Number analyzed (Participants) | 7
Participants | 2

5. Secondary Outcome: Number of Participants With Hgb in the Target Range at Week 16
Description: The number of participants with Hgb in the target range of 10.0 to 11.5 g/dL at Week 16 were analyzed. Participants who were available at the indicated time point were analyzed.
Time Frame: Week 16
Population: ITT population
Measure: Number; unit: Participants
Arm/Group | GSK1278863 12 mg QD
Number analyzed (Participants) | 7
Participants | 2

6. Secondary Outcome: Number of Participants Reaching Pre-defined Hgb Stopping Criteria
Description: The number of participants who reached the Hgb stopping criteria of Hgb concentration <7.5 g/dL from baseline to Week 16 were presented. Participants who were available at the indicated time point were analyzed.
Time Frame: Up to Week 16
Population: ITT population
Measure: Number; unit: Participants
Arm/Group | GSK1278863 12 mg QD
Number analyzed (Participants) | 15
Participants | 3

7. Secondary Outcome: Percent Change From Baseline in Hepcidin at Week 16
Description: Hepcidin is a regulator of iron metabolism. Baseline value for hepcidin is the pre-dose value on Day 1. Percent change was calculated as 100 multiplied by [exponential (log Week 16 value - log Baseline value) minus 1]. Participants who were available at the indicated time point were analyzed.
Time Frame: Baseline (Day 1) and Week 16
Population: ITT population
Measure: Geometric Mean (95% Confidence Interval); unit: Percent change in hepcidin
Arm/Group | GSK1278863 12 mg QD
Number analyzed (Participants) | 7
Percent change in hepcidin | 16.49 [-12.14 to 54.43]

8. Secondary Outcome: Change From Baseline in Ferritin at Week 16
Description: Baseline value for ferritin is the last pre-dose value on Day 1. Change from Baseline in ferritin was calculated as the Week 16 value minus the Baseline value. Participants who were available at the indicated time point were analyzed.
Time Frame: Baseline (Day 1) and Week 16
Population: ITT population
Measure: Mean (Standard Deviation); unit: Micrograms/Liter
Arm/Group | GSK1278863 12 mg QD
Number analyzed (Participants) | 7
Micrograms/Liter | -72.1 (134.81)

9. Secondary Outcome: Change From Baseline in Transferrin at Week 16
Description: Baseline value for transferrin is the last pre-dose value on Day 1. Change from Baseline in transferrin was calculated as the Week 16 value minus the Baseline value. Participants who were available at the indicated time point were analyzed.
Time Frame: Baseline (Day 1) and Week 16
Population: ITT population
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | GSK1278863 12 mg QD
Number analyzed (Participants) | 7
Percent change | 0.080 (0.2332)

10. Secondary Outcome: Percent Change From Baseline in Transferrin Saturation at Week 16
Description: Transferrin saturation is measured in percentage, it is the ratio of serum iron and total iron-binding capacity, multiplied by 100. Baseline value for transferrin saturation is the pre-dose value on Day 1. Percent change is 100 times [exponential (log Week 16 value minus log Baseline value) -1]. Participants who were available at the indicated time point were analyzed.
Time Frame: Baseline (Day 1) and Week 16
Population: ITT population
Measure: Geometric Mean (95% Confidence Interval); unit: Percent change in transferrin
Arm/Group | GSK1278863 12 mg QD
Number analyzed (Participants) | 7
Percent change in transferrin | 18.5 [-21.4 to 78.8]

11. Secondary Outcome: Change From Baseline in Total Iron at Week 16
Description: Baseline value for total iron is the last pre-dose value on Day 1. Change from Baseline in total iron was calculated as the Week 16 value minus the Baseline value. Data has been presented for only those participants who were available at indicated time points.
Time Frame: Baseline (Day 1) and Week 16
Population: ITT population
Measure: Number; unit: Micromoles (µmol)/L
Arm/Group | GSK1278863 12 mg QD
Number analyzed (Participants) | 7
Micromoles (µmol)/L
  Participant 1 | 4
  Participant 2 | 21
  Participant 3 | -3
  Participant 4 | 3
  Participant 5 | 2
  Participant 6 | 5
  Participant 7 | -5

12. Secondary Outcome: Change From Baseline in Total Iron Binding Capacity (TIBC) at Week 16
Description: Total iron-binding capacity is a medical laboratory test that measures the blood's capacity to bind iron with transferrin. Baseline value for total iron binding capacity is the last pre-dose value on Day 1. Change from Baseline in total iron binding capacity was calculated as the Week 16 value minus the Baseline value. Data has been presented for only those participants who were available at indicated time points.
Time Frame: Baseline (Day 1) and Week 16
Population: ITT population
Measure: Number; unit: µmol/ L
Arm/Group | GSK1278863 12 mg QD
Number analyzed (Participants) | 7
µmol/ L
  Participant 1 | 14
  Participant 2 | 12
  Participant 3 | -6
  Participant 4 | -1
  Participant 5 | 6
  Participant 6 | -4
  Participant 7 | 8

13. Secondary Outcome: Reticulocyte Hgb Content (CHr) at Week 16
Description: Data has been presented for only those participants who were available at indicated timepoints
Time Frame: Week 16
Population: Safety population consisted of all participants who received at least one dose of study drug
Measure: Number; unit: Picogram (pg)
Arm/Group | GSK1278863 12 mg QD
Number analyzed (Participants) | 7
Picogram (pg)
  Participant 1 | 38.80
  Participant 2 | 31.50
  Participant 3 | 32.80
  Participant 4 | 30.20
  Participant 5 | 31.70
  Participant 6 | 30.10
  Participant 7 | 34.30

14. Secondary Outcome: Mean Corpuscular Volume (MCV) at Week 16
Description: Data has been presented for only those participants who were available at indicated time points.
Time Frame: Week 16
Population: Safety population
Measure: Number; unit: Femtoliter (fL)
Arm/Group | GSK1278863 12 mg QD
Number analyzed (Participants) | 7
Femtoliter (fL)
  Participant 1 | 124.00
  Participant 2 | 99.00
  Participant 3 | 97.00
  Participant 4 | 101.00
  Participant 5 | 94.00
  Participant 6 | 97.00
  Participant 7 | 106.00

15. Secondary Outcome: Mean Corpuscular Hemoglobin (MCH) at Week 16
Description: Data has been presented for only those participants who were available at indicated time points.
Time Frame: Week 16
Population: Safety population
Measure: Number; unit: pg
Arm/Group | GSK1278863 12 mg QD
Number analyzed (Participants) | 7
pg
  Participant 1 | 39.80
  Participant 2 | 31.30
  Participant 3 | 31.70
  Participant 4 | 31.60
  Participant 5 | 30.90
  Participant 6 | 30.70
  Participant 7 | 35.70

16. Secondary Outcome: Change From Baseline in Hematocrit at Week 16
Description: Hematocrit is the ratio of the volume of red blood cells to the total volume of blood. Baseline value for hematocrit is the pre-dose value on Day 1. Change from Baseline in hematocrit was calculated as the Week 16 value minus the Baseline value. Data has been presented for only those participants who were available at indicated time points.
Time Frame: Baseline (Day 1) and Week 16
Population: ITT population
Measure: Number; unit: Fraction of 1
Arm/Group | GSK1278863 12 mg QD
Number analyzed (Participants) | 7
Fraction of 1
  Participant 1 | -0.025
  Participant 2 | 0.067
  Participant 3 | -0.015
  Participant 4 | 0.043
  Participant 5 | -0.016
  Participant 6 | 0.004
  Participant 7 | -0.089

17. Secondary Outcome: Change From Baseline in Red Blood Cell (RBC) at Week 16
Description: Baseline value for RBC (or erythrocytes) is the last pre-dose value on Day 1. Change from Baseline in red blood cells was calculated as the Week 16 value minus the Baseline value. Data has been presented for only those participants who were available at indicated time points
Time Frame: Baseline (Day 1) and Week 16
Population: ITT population
Measure: Number; unit: 10^12/L
Arm/Group | GSK1278863 12 mg QD
Number analyzed (Participants) | 7
10^12/L
  Participant 1 | -0.3
  Participant 2 | 0.7
  Participant 3 | -0.1
  Participant 4 | 0.3
  Participant 5 | -0.1
  Participant 6 | 0.2
  Participant 7 | -0.7

18. Secondary Outcome: Change From Baseline in Reticulocyte Number at Week 16
Description: Baseline value for reticulocyte number is the pre-dose value on Day 1. Change from Baseline in reticulocyte number was calculated as the Week 16 value minus the Baseline value. Data has been presented for only those participants who were available at indicated time points.
Time Frame: Baseline (Day 1) and Week 16
Population: ITT population
Measure: Number; unit: 10^12/L
Arm/Group | GSK1278863 12 mg QD
Number analyzed (Participants) | 7
10^12/L
  Participant 1 | 0.0003
  Participant 2 | 0.0043
  Participant 3 | -0.0174
  Participant 4 | -0.0139
  Participant 5 | -0.0201
  Participant 6 | -0.0458
  Participant 7 | -0.0006

19. Secondary Outcome: Maximum Observed Percent Change From Baseline in Vascular Endothelial Growth Factor (VEGF)
Description: Blood samples were collected on Day 1 (pre-dose), Week 4 (6-12 hours post-dose, then 1, 2 and 3 hours after first sample), Week 8 (pre-dose), Week 12 (pre-dose and 3 hour post-dose) and Week 16 (pre-dose) for VEGF measurement. The maximum observed percent change from Baseline in VEGF in the subjects was reported. Baseline value for VEGF is the last pre-dose value on Day 1. Percent change was calculated as 100 multiplied by exponential (log observed maximum value minus log Baseline value) minus 1. Participants who were available at the indicated time point were analyzed.
Time Frame: Baseline (Day 1) to Week 16
Population: ITT population
Measure: Geometric Mean (95% Confidence Interval); unit: Percent change
Arm/Group | GSK1278863 12 mg QD
Number analyzed (Participants) | 13
Percent change | 58.72 [35.56 to 85.84]

20. Secondary Outcome: Maximum Observed Change From Baseline in Erythropoietin (EPO)
Description: Blood samples were collected on Day 1 (pre-dose), Week 4 (6-12 hours post-dose, then 1, 2 and 3 hours after first sample), Week 8 (pre-dose), Week 12 (pre-dose and 3 hour post-dose) and Week 16 (pre-dose) for EPO measurement. The maximum observed change from baseline in EPO was reported. Baseline value for EPO is the last pre-dose value on Day 1. Change from baseline is calculated as the maximum observed value minus the baseline value. Participants who were available at the indicated time point were analyzed.
Time Frame: Baseline (Day 1) to Week 16
Population: ITT population
Measure: Mean (Standard Deviation); unit: international units(IU)/Liter (L)
Arm/Group | GSK1278863 12 mg QD
Number analyzed (Participants) | 13
international units(IU)/Liter (L) | 253.07 (526.670)

21. Secondary Outcome: Final Dose of GSK1278863
Description: For the first 4 weeks, subjects received 12mg QD of GSK1278863 with dose decrease permitted at Week 2. After 4 weeks of treatment with GSK1278863, need for dose adjustment was evaluated at visits 4, 8 and 12, to maintain hemoglobin within the target range. Target range was defined as: Hgb Criteria of 10.0 to 11.5 g/dL. Data has been presented for only those participants who were available at indicated time points.
Time Frame: Up to 16 Weeks
Population: ITT population
Measure: Number; unit: mg
Arm/Group | GSK1278863 12 mg QD
Number analyzed (Participants) | 15
mg
  Participant 1 | 25
  Participant 2 | 12
  Participant 3 | 25
  Participant 4 | 8
  Participant 5 | 12
  Participant 6 | 15
  Participant 7 | 10
  Participant 8 | 12
  Participant 9 | 0
  Participant 10 | 12
  Participant 11 | 12
  Participant 12 | 15
  Participant 13 | 15
  Participant 14 | 15
  Participant 15 | 25

22. Secondary Outcome: Plasma Concentrations of GSK1278863 and Its Metabolites at the Indicated Time Points
Description: Blood samples were collected for individual plasma GSK1278863and metabolite (GSK2391220, GSK2499166, GSK2531403, GSK2531400, GSK2531399, and GSK2531398) concentrations measurement on Day (D) 1 (pre-dose [PrD]), at Week (W) 4 (6-12, 7-13, 8-14, and 9-15 hour [hr] post-dose [PoD), and at W12 (PrD, 1, 2, and 3 hour PoD). Pharmacokinetic population: All participants from whom a PK sample has been obtained and analyzed.
Time Frame: Day 1, Week 4 and Week 12
Population: Pharmacokinetic population
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | GSK1278863 12 mg QD
Number analyzed (Participants) | 15
ng/mL
  GSK1278863, D1, PrD, n=15 | 0 (0)
  GSK1278863, W4, 6-12 hr PoD, n=13 | 64.8 (166.48)
  GSK1278863, W4, 7-13 hr PoD, n=13 | 88.6 (213.55)
  GSK1278863, W4, 8-14 hr PoD, n=13 | 79 (204.25)
  GSK1278863, W4, 9-15 hr PoD, n=13 | 67.4 (186.84)
  GSK1278863, W12, PrD, n=8 | 18 (34.15)
  GSK1278863, W12, 0.5-1 hr PoD, n=8 | 125 (186.65)
  GSK1278863, W12, 2 hr PoD, n=8 | 103.7 (140.78)
  GSK1278863, W12, 3 hr PoD, n=8 | 40.6 (32.53)
  GSK2391220, D1, PrD, n=15 | 0 (0)
  GSK2391220, W4, 6-12 hr PoD, n=13 | 41.3 (19.16)
  GSK2391220, W4, 7-13 hr PoD, n=13 | 22.6 (10)
  GSK2391220, W4, 8-14 hr PoD, n=13 | 16.7 (8.03)
  GSK2391220, W4, 9-15 hr PoD, n=13 | 12.9 (6.95)
  GSK2391220, W12, PrD, n=8 | 25.9 (22.79)
  GSK2391220, W12, 0.5-1 hr PoD, n=8 | 24.9 (21.63)
  GSK2391220, W12, 2 hr PoD, n=8 | 23.7 (19.94)
  GSK2391220, W12, 3 hr PoD, n=8 | 18 (13.43)
  GSK2487818, D1, PrD, n=15 | 0 (0)
  GSK2487818, W4, 6-12 hr PoD, n=13 | 15.8 (11.02)
  GSK2487818, W4, 7-13 hr PoD, n=13 | 9.3 (6.1)
  GSK2487818, W4, 8-14 hr PoD, n=13 | 7.2 (4.96)
  GSK2487818, W4, 9-15 hr PoD, n=13 | 5.8 (4.97)
  GSK2487818, W12, PrD, n=8 | 6.5 (9.01)
  GSK2487818, W12, 0.5-1 hr PoD, n=8 | 10.6 (10.87)
  GSK2487818, W12, 2 hr PoD, n=8 | 15.6 (19.22)
  GSK2487818, W12, 3 hr PoD, n=8 | 11.6 (11.17)
  GSK2506102, D1, PrD, n=15 | 0 (0)
  GSK2506102, W4, 6-12 hr PoD, n=13 | 13.6 (6.55)
  GSK2506102, W4, 7-13 hr PoD, n=13 | 7.5 (3.34)
  GSK2506102, W4, 8-14 hr PoD, n=13 | 5.6 (2.6)
  GSK2506102, W4, 9-15 hr PoD, n=13 | 4.3 (2.24)
  GSK2506102, W12, PrD, n=8 | 10 (7.54)
  GSK2506102, W12, 0.5-1 hr PoD, n=8 | 7.9 (6.53)
  GSK2506102, W12, 2 hr PoD, n=8 | 6.3 (4.14)
  GSK2506102, W12, 3 hr PoD, n=8 | 4.9 (3.2)
  GSK2531398, D1, PrD, n=15 | 0 (0)
  GSK2531398, W4, 6-12 hr PoD, n=13 | 16.6 (9.12)
  GSK2531398, W4, 7-13 hr PoD, n=13 | 9.4 (4.98)
  GSK2531398, W4, 8-14 hr PoD, n=13 | 7.1 (4.04)
  GSK2531398, W4, 9-15 hr PoD, n=13 | 5.6 (3.5)
  GSK2531398, W12, PrD, n=8 | 8.2 (7.78)
  GSK2531398, W12, 0.5-1 hr PoD, n=8 | 8.5 (7.57)
  GSK2531398, W12, 2 hr PoD, n=8 | 9.3 (8.71)
  GSK2531398, W12, 3 hr PoD, n=8 | 7.3 (5.75)
  GSK2531401, D1, PrD, n=15 | 0 (0)
  GSK2531401, W4, 6-12 hr PoD, n=13 | 28.4 (11.94)
  GSK2531401, W4, 7-13 hr PoD, n=13 | 15.6 (5.64)
  GSK2531401, W4, 8-14 hr PoD, n=13 | 11.6 (4.43)
  GSK2531401, W4, 9-15 hr PoD, n=13 | 8.7 (3.22)
  GSK2531401, W12, PrD, n=8 | 27.8 (22.34)
  GSK2531401, W12, 0.5-1 hr PoD, n=8 | 21 (19.46)
  GSK2531401, W12, 2 hr PoD, n=8 | 14.6 (11.05)
  GSK2531401, W12, 3 hr PoD, n=8 | 11.2 (8.83)
  GSK2531403, D1, PrD, n=15 | 0 (0)
  GSK2531403, W4, 6-12 hr PoD, n=13 | 51.8 (22.75)
  GSK2531403, W4, 7-13 hr PoD, n=13 | 28.2 (11.85)
  GSK2531403, W4, 8-14 hr PoD, n=13 | 20.6 (9.34)
  GSK2531403, W4, 9-15 hr PoD, n=13 | 15.8 (8.07)
  GSK2531403, W12, PrD, n=8 | 35.8 (28.09)
  GSK2531403, W12, 0.5-1 hr PoD, n=8 | 30.6 (25.2)
  GSK2531403, W12, 2 hr PoD, n=8 | 25.7 (18.15)
  GSK2531403, W12, 3 hr PoD, n=8 | 19.6 (13.14)

ADVERSE EVENTS:
Time Frame: On-treatment serious adverse events (SAEs) and non-serious adverse events (AEs) were collected from the start of study treatment and until the follow up (up to 20 weeks).
Description: On-treatment SAEs and non-serious AEs were reported for the Safety population consisted of all participants who received at least one dose of study drug.
Arm/Group | GSK1278863 12 mg QD
Serious Adverse Events (participants affected / at risk) | 9/15
Other Adverse Events (participants affected / at risk) | 11/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | GSK1278863 12 mg QD (N=15)
ACUTE MYOCARDIAL INFARCTION (Cardiac disorders) | 1
ANGINA UNSTABLE (Cardiac disorders) | 1
CARDIAC ARREST (Cardiac disorders) | 1
VENTRICULAR TACHYCARDIA (Cardiac disorders) | 1
GASTROENTERITIS VIRAL (Infections and infestations) | 1
PNEUMONIA (Infections and infestations) | 1
PNEUMONIA MYCOPLASMAL (Infections and infestations) | 1
GASTROINTESTINAL STOMA COMPLICATION (Injury, poisoning and procedural complications) | 1
PROCEDURAL HAEMORRHAGE (Injury, poisoning and procedural complications) | 1
HAEMATOMA (Vascular disorders) | 1
SHOCK (Vascular disorders) | 1
LOWER GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | GSK1278863 12 mg QD (N=15)
URINARY TRACT INFECTION (Infections and infestations) | 2
GASTROENTERITIS VIRAL (Infections and infestations) | 1
INFLUENZA (Infections and infestations) | 1
PNEUMONIA (Infections and infestations) | 1
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 1
NAUSEA (Gastrointestinal disorders) | 3
VOMITING (Gastrointestinal disorders) | 1
BLOOD CALCIUM DECREASED (Investigations) | 1
BLOOD PRESSURE INCREASED (Investigations) | 1
OCCULT BLOOD POSITIVE (Investigations) | 1
FATIGUE (General disorders) | 1
PYREXIA (General disorders) | 1
ARTERIOVENOUS FISTULA SITE COMPLICATION (Injury, poisoning and procedural complications) | 1
ARTERIOVENOUS FISTULA THROMBOSIS (Injury, poisoning and procedural complications) | 1
HYPERKALAEMIA (Metabolism and nutrition disorders) | 1
MALNUTRITION (Metabolism and nutrition disorders) | 1
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 2
BRACHIOCEPHALIC VEIN STENOSIS (Vascular disorders) | 1
VENOUS STENOSIS (Vascular disorders) | 1
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 1
SINUS HEADACHE (Nervous system disorders) | 1
PRURITUS (Skin and subcutaneous tissue disorders) | 1
PRURITUS GENERALISED (Skin and subcutaneous tissue disorders) | 1

LIMITATIONS AND CAVEATS:
Due to the study terminating early, resulting in a sparse amount of data, selected parameters were not summarized.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.